CLINICAL TRIAL: NCT00018174
Title: Fluoxetine as a Quit Smoking Aid for Depression-Prone Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Spring, Bonnie - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ADRD-011-97S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Smoking
Keywords: Depression; Fluoxetine; Nicotine dependence
MeSH Terms: conditions — Depression; Smoking; Tobacco Use Disorder | interventions — Fluoxetine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fluoxetine; Behavioral: Behavioral group smoking cessation treatment
- 2 (Placebo Comparator)
  Interventions: Behavioral: Behavioral group smoking cessation treatment; Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine
  Arms: 1
Behavioral: Behavioral group smoking cessation treatment
Drug: Placebo
  Arms: 2

SUMMARY:
This project is a treatment-matching study to test whether adding antidepressant pharmacotherapy to behavioral cessation treatment improves the depression-prone smoker's ability to quit, while not undermining cessation goals for the smoker who lacks a history of depression. The study target is to randomize 120 smokers with a prior history of depression and 120 smokers who lack such a history to a double-blind treatment with either 60 mg fluoxetine or placebo, while they undergo cognitive behavioral treatment to quit smoking.

DETAILED DESCRIPTION:
The aim of this research is to examine whether adding antidepressant pharmacotherapy to behavioral cessation treatment improves the depression-prone smoker's ability to quit, while not undermining cessation for the smoker who lacks a history of depression, by randomizing smokers both with and without such a history to double-blind treatment with either 60 mg fluoxetine or placebo. The primary Depressive Episode Hypothesis states that the stress of quitting smoking and the biological challenge of nicotine withdrawal trigger a depressive episode in vulnerable individuals. To the extent that episode onset can be prevented by prophylactic administration of antidepressant pharmacotherapy, smokers with a history of depression will show significantly higher abstinence rates when treated with fluoxetine than placebo, whereas no drug effect will be evident for history negative smokers who lack the depressive diathesis. An alternative generalized withdrawal hypothesis construes post-cessation dysphoria as one general manifestation of a nicotine withdrawal syndrome that occurs independently of depressive vulnerability, and predicts that fluoxetine, as compared to placebo, will uniformly improve cessation outcomes, regardless of whether smokers possess the diathesis for depression. Over period of four years, the study hopes to randomize 120 smokers with a history of depression and 120 smokers who lack such a history to double-blind treatment with either 60 mg fluoxetine or placebo, while they undergo group cognitive behavioral treatment to quit smoking. To allow plasma drug levels to stabilize before quitting smoking, drug or placebo treatment begins 3 weeks before quitting smoking and continues for an additional 8 weeks following the quit date. Participants will be followed up monthly for 4 months after the end of treatment in order to assess the main study outcome; abstinence from smoking 6 months after the quit date.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 144 smokers who have experienced at least one episode of major depressive disorder and 206 smokers who lack a lifetime history of major depressive disorder.
* None will currently meet diagnostic criteria for major depression, nor will they have met criteria in the past 6 months.
* All will be male and female community members between the ages of 18 and 65 who have smoker at least 10 cigarettes a day for the past year.

Exclusion Criteria:

Subjects may not enter the trial if they:

1. have taken monoamine oxidase inhibitors, antidepressants, anti-anxiety agents, lithium, tryptophan or phenothiazines within the past month;
2. are being treated for hypertension with guanethidine, reserpine, thiazide diuretics, beta blockers, or clonidine;
3. are taking Type IC antiarrhythmics (e.g., propafenone and flecanide) or a highly protein-bound drug (e.g., warfarin, digitoxin);
4. have a medically unstable condition or had a major health event in the past 6 months (e.g., myocardial infarct or major surgery);
5. have CBC values more than 10% outside the normal limits, or liver enzymes exceeding 40% of the upper limit of normal;
6. have a history of severe allergies, multiple adverse drug reactions or known allergy to fluoxetine;
7. are actively abusing alcohol or drugs or received inpatient treatment for substance abuse within the past year;
8. are using nicotine replacements;
9. are pregnant, lactating, or of childbearing potential;
10. present current evidence of organic brain disease, definite or subclinical major depressive disorder or serious suicidal risk post-traumatic stress disorder, or premenstrual dysphoric disorder;
11. have a score greater than 14 on the 21-item Hamilton Depression Rating Scale or greater than 15 on the Beck Depression Inventory;
12. have a history of seizures, mania or hypomania, or psychosis. Individuals with bipolar disorder, PTSD, or schizophrenia will be excluded because they might respond adversely to fluoxetine.

Subjects with dysthymic disorder or anxiety disorders will be studied if their current symptoms are not sequelae of an episode of major depression. Excluding such cases would purify the sample by removing mild degrees of dysphoria, but would greatly restrict our ability to generalize any treatment implications to the current population that smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 1998-02; Primary Completion 2003-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
tobacco abstinence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Result] Spring B, Doran N, Pagoto S, McChargue D, Cook JW, Bailey K, Crayton J, Hedeker D. Fluoxetine, smoking, and history of major depression: A randomized controlled trial. J Consult Clin Psychol. 2007 Feb;75(1):85-94. doi: 10.1037/0022-006X.75.1.85. PMID 17295567
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961